CLINICAL TRIAL: NCT05268601
Title: COVID-19 and Disease Progression to the Severe Form: a Multicentre Observational Study on the Use of Monoclonal Antibodies Against SARS-CoV-2 in Outpatients and Inpatients
Brief Title: COVID-19 and Disease Progression to the Severe Form: a Study on the Use of Monoclonal Antibodies Against SARS-CoV-2
Acronym: CONDIVIDIAMO
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Paolo Bonfanti, Director of Infectious Diseases Department, University of Milano Bicocca
Other Study IDs: MABCOVID01
Record Dates: First submitted 2022-02-25; First posted 2022-03-07 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
Keywords: SARS-CoV-2 infection; Monoclonal Antibodies; Casirivimab; Imdevimab; Bamlanivimab; Etesevimab; Sotrovimab
MeSH Terms: conditions — COVID-19 | interventions — bamlanivimab; bamlanivimab and etesevimab drug combination; casirivimab and imdevimab drug combination; sotrovimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Bamlanivimab — Administration of monoclonal antibody against SARS-CoV-2
Drug: Bamlanivimab and Etesevimab Drug Combination — Combined administration of monoclonal antibodies against SARS-CoV-2
Drug: Casirivimab and Imdevimab Drug Combination — Combined administration of monoclonal antibodies against SARS-CoV-2
Drug: Sotrovimab — Administration of monoclonal antibody against SARS-CoV-2

SUMMARY:
This is a national multicentre observational study with retrospective and prospective data collection to assess the time to hospitalisation of patients with a confirmed diagnosis of SARS-CoV-2 infection receiving treatment with anti-SARS-CoV-2 monoclonal antibodies.

The subjects enrolled will be patients with early infection of SARS-CoV-2, paucisymptomatic, with risk factors for evolution to the severe form (according to AIFA criteria). Also, hospitalised subjects will be enrolled to receive SARS-CoV-2 monoclonal antibodies because of negative serology (according to AIFA criteria).

It is estimated to enrol about 1000 subjects.

Patients will be evaluated at enrollment and 28 days following administration to collect data on symptoms, possible hospitalization and final clinical outcome (alive with symptoms, alive without symptoms, alive with symptoms and hospitalized or deceased).

Data will be collected using a dedicated electronic Case Report Form (eCRF).

ELIGIBILITY:
Inclusion Criteria:

* >/= 18 years
* Confirmed diagnosis of SARS-CoV-2 infection
* Having received or receiving any anti-SARS-CoV-2 monoclonal antibody (or combination of monoclonal antibodies) prescribed through the AIFA registry
* Signature of informed consent (for subjects enrolled in the prospective part)

Exclusion Criteria:

* Absence of criteria for prescribing monoclonal antibodies as determined by AIFA
* Patients already hospitalised for non-COVID reason at the time of monoclonal antibody administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with early infection of SARS-CoV-2, paucisymptomatic, with risk factors for evolution to the severe form (according to AIFA criteria), who receive anti-SARS-CoV-2 monoclonal antibodies.
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Estimating the time to hospitalisation of patients with a confirmed diagnosis of SARS-CoV-2 infection receiving treatment with anti-SARS-CoV-2 monoclonal antibodies up to 30 days | 0-30 days

SECONDARY OUTCOMES:
Estimating the COVID-19 lethality rate in patients receiving monoclonal antibodies (mAb) at 30 days. | 0-30 days
Describing the evolution of COVID-19 symptoms in patients receiving mAb up to 30 days | 0-30 days
Identifying possible predictive factors of hospitalisation | 0-30 days
Describing the clinical progression of patients receiving casirivimab/imdevimab while hospitalized up to 30 days | 0-30 days

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bonfanti, MD, Principal Investigator — Asst-Monza Ospedale San Gerardo
Locations (1):
- Asst-Monza Ospedale San Gerardo, Monza, Lombardy, Italy